CLINICAL TRIAL: NCT01666158
Title: Prehabilitation to Enhance Postoperative Functional Capacity Following Esophageal Resection
Brief Title: Prehabilitation for Esophageal Resection Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franco Carli (Other)
Responsible Party: Sponsor-Investigator, Franco Carli, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-171-SDR
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2016-09

CONDITIONS: Esophageal Cancer; Surgery
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Active Comparator): Patients in this group will follow standard MUHC protocol of nutritional counseling and supplementation as needed in order to maintain caloric and protein requirements in the preoperative period. Additionally, these patients will be given a specific physical exercise program before and after surgery by kinesiologist.
  Interventions: Behavioral: Exercise
- Standard nutrition counselling (No Intervention): Patients in this group will follow standard MUHC protocol of nutritional counseling and supplementation as needed in order to maintain caloric and protein requirements in the preoperative period. This group will receive general instructions on exercises (breathing, ankle rotation) to be done during hospital stay by kinesiologist.

INTERVENTIONS:
Behavioral: Exercise — The exercise component will consist of 20 min of general exercise training, 3 days per week, alternating between aerobic and resistance training. The exercise program will be individualized based upon the baseline fitness test (according to the American College of Sport Medicine, ACMS, standard) and will include: a 5 min warm-up, either 25 min of aerobic exercise (starting at 30- 40 of heart rate reserve, HRR), or 25 min of resistance training (5 exercises targeting major muscle groups performed at an intensity of 8-12 repetition maximum), and a 5 min cool-down.
  Arms: Exercise

SUMMARY:
Consenting patients scheduled for esophageal resection surgery will be randomized to receive standard nutrition counseling (including nutritional supplements as needed) or standard nutrition counseling and exercise 4 weeks before surgery and 8 weeks after surgery.

It is hypothesized that, compared with the group receiving nutrition alone, the addition of physical exercise to nutrition starting before surgery and continuing for 8 weeks after surgery will have a significantly greater impact on functional walking capacity during the prehabilitation period and during the postoperative period, and on the incidence of postoperative pulmonary complications.

DETAILED DESCRIPTION:
A randomized controlled study in patients undergoing esophageal resection for cancer to determine the impact of multimodal prehabilitation on functional exercise capacity and postoperative pulmonary complications. Patients who accept to be enrolled in the study will be randomized to receive either a standard nutritional intervention (including supplements as needed) as per current institution policy or standard nutritional intervention (including supplements as needed) combined with a physical exercise program before and after surgery.

Specific aims

The aims of this research project are the following:

1. To determine the extent in which a multimodal prehabilitation regimen optimizes functional recovery in patients suffering from esophageal cancer and the incidence of postoperative pulmonary complications.
2. To understand further which measures of immediate surgical recovery are sensitive to prehabilitation interventions, and predict change in later outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* referred electively for resection of malignant esophageal lesion

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) health status class 4-5
* Dementia and psychosis
* Disabling orthopedic and neuromuscular disease
* Severe cardiac abnormalities
* Severe end-organ disease such as cardiac failure (New York Heart Association classes I-IV)
* COPD
* renal failure (creatinine > 1.5 mg/dl, and hepatic failure ALT and AST >50% over the normal range)
* Morbid obesity (BMI >30)
* Anemia (hematocrit < 30 %, haemoglobin <10g/dl, albumin < 25mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
6 minute walk test (6MWT) | up to 8 weeks after surgery
  The 6MWT evaluates the ability of an individual to maintain a moderate level of physical activity over a time period reflective of the activities of daily living. Subjects are instructed to walk back and forth, in a 20 m stretch of hallway, for six minutes, at a pace that would make them tired by the end of the walk; encouragement and feedback are given according to published guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, M.D., Principal Investigator — Montreal University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Derived] Minnella EM, Awasthi R, Loiselle SE, Agnihotram RV, Ferri LE, Carli F. Effect of Exercise and Nutrition Prehabilitation on Functional Capacity in Esophagogastric Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2018 Dec 1;153(12):1081-1089. doi: 10.1001/jamasurg.2018.1645. PMID 30193337